CLINICAL TRIAL: NCT00936247
Title: Prospective, Controlled, Single-blind, Bicentric, Randomized Study on the Safety of HES 130/0.42 Combined With a Bal. Electr. Sol. vs 5% Albumin Comb. With an Unbal. Electr. Sol. (NaCl 0.9%) in Pat. With Compensated Renal Failure
Brief Title: Tetraspan 6 Percent (%) Combined With Sterofundin ISO Versus Albumin 5 Percent (%) Combined With Sodium Chloride (NaCL)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: organizational reasons at sites: low recruitment
Sponsor: B. Braun Melsungen AG (Industry)
Responsible Party: Dr. Simone Arnold, B. Braun Melsungen AG
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HC-G-H-0514
Record Dates: First submitted 2009-07-08; First posted 2009-07-09 (Estimated); Last update posted 2010-09-28 (Estimated); Status verified 2010-09

CONDITIONS: Renal Insufficiency
MeSH Terms: conditions — Renal Insufficiency | interventions — Albumins

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): HES 130/0.42 + Sterofundin ISO
  Interventions: Drug: HES 130/0.42 + electrolyte solution
- 2 (Active Comparator): Albumin + NaCl 0.9%
  Interventions: Drug: Albumin + electrolyte solution

INTERVENTIONS:
Drug: HES 130/0.42 + electrolyte solution — Tetraspan 6% as colloid component combined with Sterofundin ISO as electrolyte component
  Arms: 1
Drug: Albumin + electrolyte solution — Albumin 5% as colloid component and NaCl 0.9% as electrolyte component
  Arms: 2

SUMMARY:
This investigational study will investigate two different volume replacement regimes in patients suffering from compromised renal function.

ELIGIBILITY:
Inclusion:

* male or female patients
* ≥ 50 years of age;
* patients with compromised renal function, i.e. serum creatinine between 1.5 mg/dl and 3.0 mg/dl;
* patients scheduled for elective intervention;
* patients with an estimated intraoperative volume need of at least 1 l colloids;
* provision of voluntary informed consent to participate in the study, following a full explanation of the nature and purpose of the study, by signing the informed consent form approved by the Institutional Ethics Committee (IEC) prior to all evaluations

Exclusion:

* patients of ASA-class > III;
* patients with daily urine output < 1 l;
* patients on haemodialysis;
* patients receiving HES during the last 48 hours before first infusion of the investigational products;
* patients suffering from coagulation disorders (i.e. PTT > 60 sec);
* patients with a hemoglobin < 9 g/dl;
* patients with known hypersensitivity to HES, albumin or any of the excipients;
* patients suffering from contraindications of the investigational products (i.e. hyperhydration state including pulmonary oedema, renal failure with oliguria or anuria, intracranial haemorrhage, hyperkalaemia, severe hypernatraemia or severe hyperchloraemia, severely impaired hepatic function, congestive heart failure);
* simultaneous participation in another clinical trial; emergencies;
* patients scheduled for brain surgery;
* patients incapable to give informed consent (e.g. patients with dementia, psychiatric diseases or suffering from conditions associated with lack of consciousness)

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2009-11; Primary Completion 2010-09 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
Impact of two different volume replacement regimes on base excess in patients with reduced renal function | from pre-operative assessment until last evaluation of data i.e. 5th (hospital) and 60th postoperative day (follow-up)

SECONDARY OUTCOMES:
Renal function, hemodynamics, blood loss, amount of given blood products, electrolytes, outcome and other data like concomitant medication | inta-/postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Lücke, Prof. Dr., Principal Investigator — Klinikum Mannheim gGmbH, Klink für Anästhesiologie und Operative Intensivmedizin
Locations (2):
- Germany (2):
  - Klinik für Anästhesiologie und operative Intensivmedizin, Klinikum der Stadt Ludwigshafen, Ludwigshafen
  - Klinikum Mannheim gGmbH, Klinik für Anästhesiologie und Operative Intensivmedizin, Mannheim